CLINICAL TRIAL: NCT04923568
Title: Virtual Reality and Chronic Pain Pilot Usability Study
Brief Title: VR and Chronic Pain Pilot Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-13108
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- EaseVRx sessions (Experimental): This is a study of patients with chronic pain to identify interest in participating in a large VR trial and, for those willing to join us to test the device in person, to pilot 2 sessions of VR to assess usability and collect preliminary data on pain and mood and to obtain data on patient satisfaction with device use. The entire session will last 45 minutes to 1 hour. All patients recruited will be in the active arm; this is not a randomized pilot study.
  Interventions: Device: EaseVRx

INTERVENTIONS:
Device: EaseVRx — Participants will experience 2 sessions of the EaseVRx device for chronic pain

SUMMARY:
This is a pilot feasibility and usability study of a virtual reality device for patients with chronic pain.

DETAILED DESCRIPTION:
The investigators will conduct a study of patients with chronic pain to identify interest in participating in a large VR trial and, for those willing to join the team to test the device in person, to pilot 2 sessions of VR to assess usability and collect preliminary data on pain and mood and to obtain data on patient satisfaction with device use. Researchers expect the entire session to last 45 minutes to 1 hour.

All patients recruited will be in the active arm; this is not a randomized pilot study.

The intervention being piloted is the EaseVRx - AppliedVR, Los Angeles, CA - VR hardware and software. EaseVRx incorporates evidence-based principles of cognitive behavioral therapy, mindfulness, and pain neuroscience education into an immersive and enhanced biofeedback experience. EaseVRx includes breathing training and relaxation response exercises that activate the parasympathetic nervous system. EaseVRx was designed for at-home use and comes with a sequence of daily immersive experiences, with each VR experience being 2-16 minutes in length (average of 6 minutes). For this pilot, researchers will be doing one in-person session, using two interoceptive VR experiences (out of 56 total).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Chronic pain (using self-report) with pain intensity >=4 and confirmed by ICD-10 codes in medical record
3. Fluency in English

Exclusion Criteria:

1. Inability to give informed consent
2. Current or prior diagnosis of epilepsy, seizure disorder, dementia, migraines
3. Medical condition predisposing to nausea or dizziness
4. Hypersensitivity to flashing light or motion
5. No stereoscopic vision or severe hearing impairment
6. Injury to eyes, face, or neck that prevents use of VR headset
7. Currently pregnant, by self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
% of participants contacted that are enrolled | at study 1 day visit
  We will determine feasibility by measuring the % of participants that are contacted who are enrolled.

SECONDARY OUTCOMES:
Satisfaction with VR experience | at study 1 day visit
  We use the Global Impression of Change Scale, which is a 7 point Likert type scale, at the conclusion of the VR experience to measure patient's perceived impression of change before and after VR.
Change in Mood | at study 1 day visit
  We use the Brief Mood Introspection Scale, a 16-item scale, to measure change in mood before and after VR
Change in Pain intensity | at study 1 day visit
  We use a 1-item pain intensity score (0-10) both before and after VR

CONTACTS AND LOCATIONS:
Overall Officials: Hector R Perez, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No